CLINICAL TRIAL: NCT04431557
Title: The Electroencephalogram Analysis in the Differences Between Inhalation Anesthetic and Propofol.
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201509018RINB
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2017-07

CONDITIONS: Sevoflurane; Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will record 120 patients who received general anesthesia, their EEG data recorded from Bispectral Index (BIS) machine for emperical mode decomposition (EMD) analysis, the investigators decomposed EEG signal to different oscillations and tried to observe the differences between hypnotic medications through EEG analysis.

DETAILED DESCRIPTION:
The electroencephalography (EEG) is a noninvasive medical technique for monitoring and recording the electrical activity of brain. The Hilbert-Huang transform (HHT) was proposed to decompose EEG signal into intrinsic mode functions (IMF) which can obtain instantaneous frequency data and work well for data that is nonstationary and nonlinear.

The relationship between frontal EEG patterns and hypnotics remain poorly understood. The investigators only can tell the increase in frontal EEG power and shift power to lower frequencies during general anesthesia from publications. The investigators are going to decompose EEG with HHT and find the energy shift during general anesthesia, compare with different anesthetics.

The investigators will record 120 patients who received general anesthesia, their EEG data recorded from BIS machine for EMD analysis, the investigators decomposed EEG signal to different oscillations and tried to observe the differences between hypnotic medications through EEG analysis.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* scheduled surgery who need general anesthesia

Exclusion Criteria:

* allergy to the BIS patch
* not suitable for general anesthesia

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population was focus on the patients who need schedule general anesthesia with low anesthesia risk (ASA I-II).
Sampling Method: Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
The gamma, beta, alpha and theta power of EEG | the total duration inclusions in operation room
  We will try to observe the differences between hypnotic medications through EEG decomposed and power analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Fang Tsai, M.D., Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan